CLINICAL TRIAL: NCT07271940
Title: Full Plate Living Nutrition Education Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1466; Approval 11/20/25 (Other: UW Madison); SMPH/DOM General Internal (Other: UW Madison)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus; Pre Diabetes; Obesity
Keywords: fiber; nutrition
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full Plate Living Nutrition Education Program (Experimental)
  Interventions: Other: Full Plate Living Nutrition Education Program

INTERVENTIONS:
Other: Full Plate Living Nutrition Education Program — Participants will attend 8 sessions over 8 weeks. Participants will learn about the importance of fiber and how to add fiber to their diet.

SUMMARY:
The purpose of the research is to evaluate the acceptability and feasibility of implementing a 8-session nutritional education program in a general internal medicine clinic. This program emphasizes a fiber-rich, whole foods diet consisting of fruits, vegetables, legumes, whole grains, nuts and seeds. Such interventions can improve diabetes management and lead to weight loss. 48 participants will be enrolled and on study for approximately 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Pre-diabetes or diabetes
* Body Mass Index (BMI) 30-42
* UW Health Primary Care Physician

Exclusion Criteria:

* Pregnant
* Active cancer (treatment within one year or planning on having treatment)
* Eating Disorder (SDE Screening 2+)
* Chronic Kidney Disease (CKD) (Stage 4 or 5)
* Patient Health Questionnaire-9 (PHQ9) indicating severe depression (greater than 15)
* No PHQ9 and PHQ2 greater than 2
* General Anxiety Disorder-7 (GAD7) indicating severe anxiety (greater than 15)
* No GAD 7 and GAD2 greater than 2
* Inflammatory bowel disease (IBD)
* Irritable bowel syndrome (IBS)
* Readiness to Change less than 7
* Confidence to Change less than 7
* Lack of transportation
* Non-English Speaking
* No control over food environment
* No access to laptop, desktop computer, or tablet
* No email or text message access
* Unwilling to participate in a shared medical visit
* Unable to attend one of the four concurrent shared medical visit session cohorts
* For those on insulin, no access to finger-prick blood glucose meter or continuous glucose monitor

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Participant Weight | retrospectively from 2 years prior to enrollment and up to 20 weeks on study (3 month follow up)

SECONDARY OUTCOMES:
Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) | baseline, 8 weeks, 20 weeks (3 month follow up)
  Dietary fiber (grams per day) will be measured using the Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24) which has been validated for measuring fiber intake in adults. The ASA24 is a free, web-based tool. Participants will complete the ASA24 online two times prior to the first session, 2 times prior to the last session, and 2 times 3 months after the last session.
Participant Quality of Life measured by the SF-12 score | baseline, 8 weeks, 20 weeks (3 month follow up)
  Possible scores range from 0-100 with higher scores indicating better quality of life.
Acceptability: Percent of Participants who found the intervention acceptable | Participant surveyed at the end of last session, approximately 8 weeks
  A subset of participants will be invited to complete an individual interview after the last session. The aim is to schedule 8-12 participants for interviews including both participants who completed all the sessions and those stopped attending sessions. Data will be derived from these qualitative semi-structured interviews.
Feasibility: Participant Retention Rate | baseline, 8 weeks, 20 weeks (3 month follow up)
  Feasibility will in part be measured by participant retention rate, the number of participants who complete each time point of data collection over the number of participants enrolled.
Feasibility: Participation Rate | Through enrollment (up to 3 months)
  Feasibility will in part be measured by participation rate, the number of participants enrolled over the target enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Miller, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No